CLINICAL TRIAL: NCT01002469
Title: Pilot Feasibility Study in Healthy Subjects and Healthy Asymptomatic Subjects Genetically Disposed to Urea Cycle Disorders to Evaluate the Use of 13 C Isotope Ratio Measurement
Brief Title: Study to Evaluate 13 C Isotope Ratio Measurement for Urea Cycle Capacity Assessment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cytonet GmbH & Co. KG (Industry)
Responsible Party: Heinz Kriegbaum, Cytonet GmbH & Co. KG
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CCD07
Record Dates: First submitted 2009-10-26; First posted 2009-10-27 (Estimated); Last update posted 2010-01-15 (Estimated); Status verified 2010-01

CONDITIONS: Urea Cycle Disorders
Keywords: isotope ratio measurement; urea cycle; 13C acetate; Healthy adults
MeSH Terms: conditions — Urea Cycle Disorders, Inborn | interventions — Sodium; Acetates

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- sodium [1-13C] acetate (Experimental)
  Interventions: Other: sodium [1-13C] acetate

INTERVENTIONS:
Other: sodium [1-13C] acetate

SUMMARY:
In this short-term study a method for the evaluation of the metabolic competency of the urea cycle in vivo will be assessed. In order to monitor the efficacy of new treatment options for patients with urea cycle disorders and to monitor the severity of the disease, a reliable and safe quantitative method for the measurement of the urea cycle flux is required.

Urea synthesis will be evaluated by administering sodium [1-13C]-acetate and measuring subsequent incorporation of [13C] label from Na-acetate into urea in healthy volunteers and asymptomatic subjects genetically disposed to urea cycle disorders.

ELIGIBILITY:
Inclusion Criteria:

* Group 1 + 2: Healthy subjects
* Group 3: Healthy asymptomatic subjects genetically disposed to urea cycle disorders
* All: age 18 to 50 years (adult)
* Written informed consent

Exclusion Criteria:

* Presence of acute infection
* Participation in other clinical trials within 30 days prior to inclusion
* Severe coagulopathy
* Severe systemic or chronic disease
* Pregnancy or lactation

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2009-09; Primary Completion 2009-11 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Increase of [13C]urea AUC in plasma following oral administration of [13C ]-sodium acetate over baseline

SECONDARY OUTCOMES:
Cmax of absolute [13C]urea in plasma

CONTACTS AND LOCATIONS:
Overall Officials: Doris Neuenhofer, MD, Principal Investigator — CRS Clinical Research Services Mönchengladbach GmbH
Locations (1):
- CRS Clinical Research Services Mönchengladbach GmbH, Mönchengladbach, Germany